CLINICAL TRIAL: NCT05314283
Title: A Feasibility Study Investigating the Safety, Performance and Gastrointestinal Transit of the DV3395 Device Concept in Healthy Participants.
Brief Title: A Study Investigating the Safety and Performance of DV3395, a New Concept Device for the Delivery of Medicine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DV3395-4711; U1111-1253-1898 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-03-18; First posted 2022-04-06 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers, Medical Device

STUDY DESIGN:
Intervention Model Description: Including a pilot cohort and a main cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DV3395 C1 (Experimental)
  Interventions: Device: DV3395 C1

INTERVENTIONS:
Device: DV3395 C1 — Participants will be exposed to and swallow DV3395 C1 once. The participants will stay at the clinic research center for up to 6 days .

SUMMARY:
This study investigates how safe the study device DV3395-C1 is when swallowed by healthy men and women. By the use of X-ray the device will be followed from the mouth, through the food pipe to the stomach and then into the gut. It will be checked if the device activates itself in the stomach as planned. Participants will be admitted to the clinic research center on day -1 and will receive the device on day 1 after 6 hours fast. The X-ray session will take up to 5 hours ending with administration of a small amount of contrast agent for better visualisation. The participants will stay at the clinic research center for up to 6 days until the device has been excreted. A follow-up phone call will take place 1 week after the device has been excreted.

ELIGIBILITY:
Inclusion criteria:

* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Body mass index between 18.5 and 29.9 kg/m^2 (both inclusive).

Exclusion criteria:

* Presence of any known or suspected clinically significant gastrointestinal disease or gastrointestinal disorder (including functional and structural disorders) as judged by the investigator.
* History of clinically significant gastrointestinal or abdominal surgery (including gynaecological/obstetrical and urological procedures) as judged by the investigator.
* History of radiotherapy of the neck, thorax or abdomen.
* Exposure to ionizing radiation from diagnostic or interventional procedures of greater than 0.1 mSv within 1 year prior to V2 pre-administration, a radiation burden of greater than 1.1 mSv within 2 years prior to V2 pre-administration, a radiation burden of greater than 2.1 mSv within 3 years prior to V2 pre administration, etc. (add 1 year per 1 mSv).
* Known or suspected hypersensitivity to any component of DV3395 C1 or to any iodine based contrast agent.
* Female for whom any of the below applies:

  * pregnant as determined by a positive laboratory pregnancy test at screening or at V2 pre administration
  * breast-feeding
  * of child-bearing potential and not using an adequate contraceptive method for 28 days or more prior to screening or between screening and V2 pre-administration, and not willing to maintain use of adequate contraception during the study period (adequate contraceptive measures as required by local regulation or practice)
  * wish to become pregnant within 6 months after the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | From exposure (defined as when the participant takes DV3395-C1 into his/her hand with the intention of swallowing it) to DV3395 C1 on day 1 (visit 2) to 7 days after excretion of DV3395 C1 (phone visit 3, expected between day 9 and day 12)
  Number of events

SECONDARY OUTCOMES:
Confirmed DV3395 C1 integrity upon excretion (yes/no) | On day of excretion of DV3395 C1 (visit 2, expected between day 2 and day 5)
  Count of participant
Confirmed gastric activation of DV3395 C1 (yes/no) | From administration (defined as when the participant places DV3395-C1 in his/her mouth with the intention of swallowing it) of DV3395 C1 on day 1 (visit 2) to time of last image approximately 5 hours later on day 1 (visit 2)
  Count of participant
Time to activation of DV3395 C1 | From administration (defined as when the participant places DV3395-C1 in his/her mouth with the intention of swallowing it) of DV3395 C1 on day 1 (visit 2) to time of last image approximately 5 hours later on day 1 (visit 2)
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- ICON - location Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com